CLINICAL TRIAL: NCT04520217
Title: Pilot Studies Testing Use of Topical Imipramine in Reducing Ultraviolet B Induced Microvesicle Particle Release in Photosensitive Subjects
Brief Title: Testing Use of Topical Imipramine in Reducing Ultraviolet B Induced Microvesicle Particle Release in Photosensitive Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 06919
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Photosensitivity; Microvesicle Particle
MeSH Terms: conditions — Photosensitivity Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 4% Imipramine Cream on UVB-Treated Areas (Experimental): * 2g of 4% imipramine cream will be applied to the UVB-treated areas on volar forearm and back.
  * 2g of base cream will be applied to the UVB-treated areas on volar forearm and back.
  * No cream will be applied to a UVB-treated area on the back
  Interventions: Drug: 4% Imipramine Cream; Drug: Base Cream

INTERVENTIONS:
Drug: 4% Imipramine Cream — 4% Imipramine Cream
Drug: Base Cream — Base Cream

SUMMARY:
The purpose of this study is three-fold. First, researchers will assess whether subjects who have clinically abnormal reactions to sunlight (photosensitivity) have increased levels of microvesicle particles (MVP) following ultraviolet B (UVB) treatment to localized area of skin. Second, researchers will assess if topical application of the medicine imipramine will block UVB-induced MVP release. Third, researchers will assess if the topical cream will block UVB-induced increased erythema reactions (reddening of the skin).

ELIGIBILITY:
Inclusion Criteria:

* Female and Male adult subjects age 18 to 50
* Must be able to give informed consent
* Have access to stable transportation
* All skin types on Fitzpatrick Scale (Type I-VI)
* Self-Identified photosensitivity
* Able to provide medical history and list of medications-control subjects will not be allowed to be taking a medication that is known to be photosensitizer.

Exclusion Criteria:

* Underlying diseases that could affect wound healing (e.g., uncontrolled diabetes mellitus)
* Taking medications that are known photosensitizers (e.g., doxycycline) or anti-inflammatories (e.g., NSAIDS [except for low-dose aspirin] or steroids)
* Utilizing imipramine or any other tricyclic antidepressant (oral or cream)
* Utilizing topical anti-inflammatory or systemic agents (e.g., prednisone)
* Large tattoos in the designated testing areas
* Tanning bed use within last 3 months
* Photodynamic Therapy or UVB treatments in past 3 months
* Female Subjects: pregnant or nursing
* History of abnormal scarring (i.e., keloids)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in microvesicle particle levels from baseline in clinically photosensitive subjects | 4 Hours
  This will be measured in skin biopsies obtained at 4 hours following ultraviolet B radiation fluence of 1000 J/m2.
Change in microvesicle particle levels from baseline post topical imipramine application | 4 Hours
  This will be measured in skin biopsies with topical imipramine applied. Biopsies are obtained at 4 hours following ultraviolet B radiation fluence of 1000 J/m2.
Change in skin erythema from baseline on topical imipramine treated skin | 4 Hours
  This will be measured with a mexameter at 4 hours.
Change in skin erythema from baseline on topical imipramine treated skin | 24 Hours
  This will be measured with a mexameter at 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Travers, MD, PhD, Principal Investigator — Wright State University
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT04520217/ICF_000.pdf